CLINICAL TRIAL: NCT05303129
Title: Prognostic Impact of the Neutrophil/Lymphocyte Ratio (NLR) in the Treatment of First-line Metastatic or Locally Advanced Breast Cancer Treated With CDK4/6 in
Brief Title: Prognostic Impact of the Neutrophil/Lymphocyte Ratio (NLR) in the Treatment of First-line Metastatic or Locally Advanced Breast Cancer Treated With CDK4/6 Inhibitor.
Acronym: PEPSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021-A02664-37
Record Dates: First submitted 2022-03-21; First posted 2022-03-31 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer; Metastatic Breast Cancer
Keywords: CDK4/6; lymphocyte typing; Neutrophil/Lymphocyte ratio (NLR)
MeSH Terms: conditions — Breast Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood tests (Other): Realization of 4 blood tests for Lymphocyte typing (Neutrophil/Lymphocyte ratio (NLR), CD4+ and CD8+ lymphocyte counts ), during CDK4/6 treatment :
  * before initiation of CDK4/6 treatment
  * At 3 mois after initiation of CDK4/6 treatment
  * At 6 mois after initiation of CDK4/6 treatment
  * At 12 mois after initiation of CDK4/6 treatment or at early end of study
  Interventions: Biological: Blood sampling

INTERVENTIONS:
Biological: Blood sampling — Blood sampling for Lymphocyte typing (Neutrophil/Lymphocyte ratio (NLR), CD4+ and CD8+ lymphocyte counts )

SUMMARY:
The impact of the inflammatory microenvironment in predicting the benefit of a CDK4/6 inhibitor in the treatment of locally advanced or first line metastatic breast cancer has not yet been studied.

We propose a multicenter prospective study to confirm the prognostic value of pre-therapy NLR on progression-free survival of patients initiating treatment with a CDK4/6 inhibitor combined with hormonal therapy for locally advanced or metastatic HR-pos / HER2-neg breast cancer.

We will also evaluate other markers of inflammation and their prognostic and predictive value for a better response to CDK4/6 inhibitor therapy in combination with hormone therapy in these patients.

Specific blood tests (lymphocyte typing) will be performed during treatment with CDK4/6.

DETAILED DESCRIPTION:
The impact of the inflammatory microenvironment in predicting the benefit of a CDK4/6 inhibitor in the treatment of locally advanced or first line metastatic breast cancer has not yet been studied.

We propose a multicenter prospective study to confirm the prognostic value of pre-therapy NLR on progression-free survival of patients initiating treatment with a CDK4/6 inhibitor combined with hormonal therapy for locally advanced or metastatic HR-pos / HER2-neg breast cancer.

We will also evaluate other markers of inflammation and their prognostic and predictive value for a better response to CDK4/6 inhibitor therapy in combination with hormone therapy in these patients.

Specific blood tests (lymphocyte typing) will be performed during treatment with CDK4/6.

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced or metastatic HR-positive, Her2-negative breast cancer
* Patients who are scheduled to receive first-line metastatic CDK4/6 inhibitor therapy in combination with hormone therapy as per the marketing authorization
* Patients who have not received previous anti-neoplastic therapies for metastatic or advanced disease (chemotherapy, targeted therapy or hormonal therapy). However, it will be possible to have initiated 1st line hormonal therapy within 4 to 6 weeks prior to inclusion.
* Prior radiotherapy allowed even in metastatic disease. In case of radiotherapy treatment, side effects attributable to the treatment must be resolved.
* Postmenopausal patients or patients with suppressed ovarian function
* Patient with measurable or non-measurable disease (according to RECIST v1.1 criteria)
* Adequate organ and marrow function to allow prescription of CDK 4/6 inhibitor therapy
* Age of Patient ≥ 18 years
* Willingness and ability to comply with scheduled visits, treatment plan, biologic tests and other trial procedures including assessments requested for inclusion
* Patient affiliated with a social security plan
* Informed consent signed prior to any specific study-related procedures

Exclusion Criteria:

* Men (no marketing authorization for CDK4/6 inhibitors in men in France)
* Previous systemic treatment for metastatic disease (chemotherapy, hormone therapy, etc.)
* Previous treatment with a CDK4/6 inhibitor (adjuvant or for metastatic disease)
* Locally advanced or relapsed breast cancer for which curative treatment would be considered
* Her2-positive tumor status on either the primary or relapsed tumor as defined by ASCO criteria
* Patient with advanced, symptomatic visceral extension who may be at risk for a potentially fatal short-term complication ("visceral crisis") and who requires treatment with chemotherapy
* Patients who are deprived of their liberty, under guardianship, or subject to a legal protection measure or who are unable to express their consent
* Patients who cannot undergo the trial follow-up for geographical, social or psychopathological reasons

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2022-05-27 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2024-12-17 (Actual)

PRIMARY OUTCOMES:
Progression-free survival rate | At 12 months after initiation of CDK 4/6 treatment
  Progression-free survival rate according to the Neutrophil/Lymphocyte (NLR) ratio. NLR cut-off set at 2.53

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre François Baclesse, Caen
  - Centre Henri BECQUEREL, Rouen

IPD SHARING:
Plan to Share IPD: No